CLINICAL TRIAL: NCT05289973
Title: Effect of TruNatomy and HyFlex EDM Instrumentation on Postoperative Pain in Asymptomatic Necrotic Molars.
Brief Title: Effect of TruNatomy and HyFlex EDM Instrumentation on Postoperative Pain
Acronym: TRN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora El-Sayed Khater, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRN in postoperative pain
Record Dates: First submitted 2021-12-22; First posted 2022-03-22 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: patients having mandibular molars with necrotic pulp
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TruNatomy Files (Experimental): Newly introduced endodontic file
  Interventions: Device: TruNatomy Files
- Hyflex EDM (Experimental): Endodontic file
  Interventions: Device: HyFlex EDM Files

INTERVENTIONS:
Device: TruNatomy Files — Newly introduced endodontic file with high flexibility.
  Arms: TruNatomy Files
Device: HyFlex EDM Files — Endodontic files
  Arms: Hyflex EDM

SUMMARY:
The aim of the present study is to clinically compare the incidence of postoperative pain after root canal preparation using TruNatomy system and HyFlex Electrical Discharge Machined (EDM) rotary system in asymptomatic necrotic mandibular molars.

DETAILED DESCRIPTION:
Up till now, there are no clinical studies on the effect of instrumentation using TruNatomy files on post-operative pain. Furthermore, these newly introduced files can provide more affordable means for instrumentation. Therefore, the purpose of this study is to clinically compare the effect of using TruNatomy files and HyFlex EDM files on post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 - 45 years old.
2. Males or Females.
3. Mandibular molar teeth with:

   * No pain.
   * No response to pulp testing.
   * Radiographic appearance with or without a periapical radiolucency.

Exclusion Criteria:

1. Patients with pre-operative pain.
2. Patients having significant systemic disorders.
3. Patients who are allergic to non-steroidal anti-inflammatory drugs.
4. Patients with two or more adjacent teeth requiring root canal therapy.
5. Teeth that have:

   * Vital pulp tissues.
   * Association with swelling or fistulous tract.
   * Acute or chronic peri-apical abscess.
   * Greater than grade I mobility.
   * Pocket depth greater than 5mm.
   * No possible restorability.
   * Previous endodontic treatment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain : measure pain level change from zero(no pain) pain Post-operative pain Post-operative pain | Post-operative pain measured 6, 12, 24, 48, 72 hours and 7 days post-operatively.
  The pain will be recorded according to the modified visual analogue scale. The scale consists of a line marked from 1 to 10 where 10 represent the most intense pain imaginable and the worst outcome.

SECONDARY OUTCOMES:
Number of analgesics taken by the patient after endodontic treatment | up to 7 days post-operatively
  Counting Number of analgesics taken by the patient after endodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Angie Ghoneim, PHD, Study Director — Cairo University

REFERENCES:
- [Background] Thompson SA. An overview of nickel-titanium alloys used in dentistry. Int Endod J. 2000 Jul;33(4):297-310. doi: 10.1046/j.1365-2591.2000.00339.x. PMID 11307203
- [Background] Arias A, de la Macorra JC, Hidalgo JJ, Azabal M. Predictive models of pain following root canal treatment: a prospective clinical study. Int Endod J. 2013 Aug;46(8):784-93. doi: 10.1111/iej.12059. Epub 2013 Feb 12. PMID 23402273
- [Background] Ruiz-Hubard EE, Gutmann JL, Wagner MJ. A quantitative assessment of canal debris forced periapically during root canal instrumentation using two different techniques. J Endod. 1987 Dec;13(12):554-8. doi: 10.1016/S0099-2399(87)80004-3. No abstract available. PMID 3482231